CLINICAL TRIAL: NCT05875246
Title: Stress Physiology and Intervention Feasibility Among First Responder Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Chapman University (Other)
Responsible Party: Principal Investigator, Abigail Gewirtz, Professor, Arizona State University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00017540
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Stress; Parenting

STUDY DESIGN:
Intervention Model Description: 30-day cycle involving the EMA Questions, along the micro-Intervention randomization and delivery. The application is coded to randomize each participant to one of the three intervention options. During this 30-day cycle physiological data will be collected from the Garmin Vivosmart 5 device worn by the participant and loaded into the Labfront app for storage and retrieval.
  MYAPT.MIND (Daily for 30 days)
  * Ecological Momentary Assessment (EMA) Survey Questions Set #1
  * Micro-Intervention (None, Brief Messages, MYAPT.MIND Audios)
  * Ecological Momentary Assessment (EMA) Survey Questions Set #2
  * HRV (Heart Rate Variability) via Garmin Vivosmart 5 wrist wearable
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (No Intervention): Does not receive a micro-intervention
- Group 2 (Experimental): Receives brief messages for stress reduction.
  Interventions: Behavioral: Micro-interventions
- Group 3 (Experimental): Directed to the app to listen to a stress reduction audio activity.
  Interventions: Behavioral: Micro-interventions

INTERVENTIONS:
Behavioral: Micro-interventions — Group 1: No intervention Group 2: Brief stress reduction messages Group 3: App based stress reduction audio activity
  Arms: Group 2; Group 3

SUMMARY:
The specific aims of this study are to: 1. Demonstrate the usability and acceptability of a smart watch in parents to remotely monitor stress responses or symptoms in individuals participating in prevention or treatment interventions. 2. Examine the association between heart rate variability (HRV) data and momentary self-reports of stress by parents. 3. Conduct a feasibility study to establish the effectiveness of wearables and apps to improve emotion regulation in the short term (minutes, hours) and concomitant social, emotional, and behavioral outcomes over the longer-term (weeks).

ELIGIBILITY:
Inclusion Criteria:

* Have at least one child between the ages of 4 and 13 that resides with them in states of Kentucky or Tennessee
* Be able to wear a wrist-based wearable device
* Be able to read, write, and speak in English
* Not be allergic to polycarbonate or silicone
* Have a smart phone
* Work full time (at least 30 hours/week) as a first responder OR be a co-parent (defined as living in the same home and shares parenting responsibilities) of an eligible first responder

Exclusion Criteria:

* Do not have a child in the specified age range
* Have a child in the specified age range but who does not reside with them
* Are first responders who average less than 30 hours/week
* Are not a cohabitating parent
* Are a co-parent of eligible first responders who is not participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 30 days
  HRV collected via wearables device
EMAs | 30 days
  Self-report of stress

CONTACTS AND LOCATIONS:
Overall Officials: Abi Gewirtz, PhD, Principal Investigator — Arizona State University
Locations (2):
- United States (2):
  - First Responders State Wide, Clarksville, Kentucky
  - First Responders State Wide, Charlotte, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided